CLINICAL TRIAL: NCT02959892
Title: A Phase 1, Open-Label, Positron Emission Tomography Study in Healthy Subjects to Determine the Effect of TAK-041 on Amphetamine-Induced Dopamine Release in the CNS After Single-Dose Oral Administration
Brief Title: A Single-Dose Positron Emission Tomography (PET) Study to Determine the Effect of TAK-041 on Amphetamine-Induced Dopamine Release in the Central Nervous System (CNS)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Neurocrine Biosciences (Industry)
Collaborators: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: TAK-041-1002; U1111-1184-1947 (Registry Identifier: WHO); 2016-002346-23 (EudraCT Number)
Record Dates: First submitted 2016-11-07; First posted 2016-11-09 (Estimated); Results first posted 2019-12-23 (Actual); Last update posted 2021-03-19 (Actual); Status verified 2021-03

CONDITIONS: Healthy Volunteers
Keywords: Drug therapy
MeSH Terms: interventions — Amphetamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TAK-041 20 mg (Experimental): [11C] PHNO 180 megabecquerel (MBq), injection, intravenously, prior to positron emission tomography (PET) scan on Day 1, followed by amphetamine (AMPH) 0.5 milligram per kilogram (mg/kg), tablet, orally, once and [11C] PHNO 180 MBq, injection, intravenously, prior to PET scan post-AMPH dose on Day 2 of Confinement Period 1, followed by a 5 to 45 days of interval period, further followed by TAK-041 20 mg, suspension, orally, once, followed by AMPH 0.5 mg, tablet, orally, once and [11C] PHNO 180 MBq, injection, intravenously, prior to PET scan post-AMPH dose on Day 1 of Confinement Period 2.
  Interventions: Drug: Amphetamine; Drug: TAK -041; Drug: [11C] (+)-4-propyl-(+)-4-propyl-9-hydroxynaphthoxazine (PHNO)
- TAK-041 40 mg (Experimental): [11C] PHNO 180 MBq, injection, intravenously, prior to PET scan on Day 1, followed by AMPH 0.5 mg/kg, tablet, orally, once and [11C] PHNO 180 MBq, injection, intravenously, prior to PET scan post-AMPH dose on Day 2 of Confinement Period 1, followed by a 5 to 45 days of interval period, further followed by TAK-041 40 mg, suspension, orally, once, followed by AMPH 0.5 mg, tablet, orally, once and [11C] PHNO 180 MBq, injection, intravenously, prior to PET scan post-AMPH dose on Day 1 of Confinement Period 2.
  Interventions: Drug: Amphetamine; Drug: TAK -041; Drug: [11C] (+)-4-propyl-(+)-4-propyl-9-hydroxynaphthoxazine (PHNO)

INTERVENTIONS:
Drug: Amphetamine — Amphetamine tablets.
Drug: TAK -041 — TAK-041 oral suspension.
Drug: [11C] (+)-4-propyl-(+)-4-propyl-9-hydroxynaphthoxazine (PHNO) — [11C]PHNO injection.

SUMMARY:
The purpose of this study is to determine brain penetration of single oral doses of TAK-041 and its effects on amphetamine-induced dopamine release in the Central Nervous System (CNS).

DETAILED DESCRIPTION:
The drug being tested in this study is called TAK-041. This study will look at brain penetration of single oral doses of TAK-041 and its effects on amphetamine-induced dopamine release in the CNS.

The study will enroll participants until 12 evaluable participants complete all study procedures. The first 4 participants enrolled in this study will receive a dose of 20 mg TAK-041 and 0.50 milligram per kilogram (mg/kg) dose of amphetamine. The dose for subsequent participants will be determined based on the results of amphetamine-induced dopamine release in the first 4 participants (5 to 40 for TAK-041 and 0.25 or 0.50 mg/kg for the amphetamine).

This single-center trial will be conducted in the United Kingdom. The overall time to participate in this study is approximately 92 days. Participants will remain confined to the clinic for 3 to 4 days during 2 confinement periods. Participants will make monthly visits during Days 8-64 and a final visit 30 days later.

ELIGIBILITY:
Inclusion Criteria:

1. Is in good health as determined by physical examination, electrocardiogram (ECG), and laboratory evaluations.
2. Weighs at least 45 kilogram (kg) and has a body mass index (BMI) from 18.0 to 30.0 kilogram per square meter (kg/m^2), inclusive, at Screening.

Exclusion Criteria:

1. Has a history of drug abuse (defined as any illicit drug use) or a history of alcohol abuse (defined as regular consumption of more than 21 units per week) within 1 year prior to the Screening Visit or is unwilling to agree to abstain from alcohol and drugs throughout the study. One unit is equivalent to 8 grams of pure alcohol, which is equivalent to 10 milliliter (mL) of pure ethanol (alcohol) or approximately a half-pint of beer, 1 measure of spirits, or 1 glass of wine.
2. Has used nicotine-containing products (including but not limited to cigarettes, pipes, cigars, chewing tobacco, nicotine patch or nicotine gum) within 28 days prior to Check-in on Day -1. Cotinine test is positive at Screening or Check-in (Day -1).
3. Has poor peripheral venous access.
4. Has donated or lost 450 mL or more of his blood volume (including plasmapheresis), or had a transfusion of any blood product within 90 days prior to Confinement Period 1.
5. Has had previous research-related exposure to ionizing radiation such that, in combination with the exposure from this study, their exposure will be greater than (>)10 millisievert (mSv) for the previous year.
6. Has a contraindication to magnetic resonance imaging (MRI) based on the standard MRI screening questionnaire. Contraindications include ferromagnetic foreign bodies (example, shrapnel, ferromagnetic fragments in the orbital area), certain implanted medical devices (example, aneurysm clips, cardiac pacemakers), or claustrophobia.
7. Has findings on the screening brain MRI scan that will potentially compromise participant safety or the scientific integrity of the study data if the participant were to participate in this study.

Ages: 20 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 12 (Actual)
Dates: Start 2016-12-05 (Actual); Primary Completion 2017-05-30 (Actual); Study Completion 2017-08-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Takeda
Locations (1):
- Hammersmith Medicines Research, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Takeda makes patient-level, de-identified data sets and associated documents available after applicable marketing approvals and commercial availability have been received, an opportunity for the primary publication of the research has been allowed, and other criteria have been met as set forth in Takeda's Data Sharing Policy (see www.TakedaClinicalTrials.com/Approach for details). To obtain access, researchers must submit a legitimate academic research proposal for adjudication by an independent review panel, who will review the scientific merit of the research and the requestor's qualifications and conflict of interest that can result in potential bias. Once approved, qualified researchers who sign a data sharing agreement are provided access to these data in a secure research environment.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 1 investigative site in United Kingdom from 05 December 2016 to 23 August 2017.
Pre-assignment Details: Healthy participants were enrolled in this study to receive TAK-041 in one of the 2 treatment groups: TAK-041 20 milligram (mg) or TAK-041 40 mg.
Groups:
- TAK-041 20 mg: [11C] (+)-4-propyl-(+)-4-propyl-9-hydroxynaphthoxazine (PHNO) 180 megabecquerel (MBq), injection, intravenously, prior to positron emission tomography (PET) scan on Day 1, followed by amphetamine (AMPH) 0.5 milligram per kilogram (mg/kg), tablet, orally, once and [11C] PHNO 180 MBq, injection, intravenously, prior to PET scan post-AMPH dose on Day 2 of Confinement Period 1, followed by a 5 to 45 days of interval period, further followed by TAK-041 20 mg, suspension, orally, once, followed by AMPH 0.5 mg, tablet, orally, once and [11C] PHNO 180 MBq, injection, intravenously, prior to PET scan post-AMPH dose on Day 1 of Confinement Period 2.
Period: Overall Study
Arm/Group | TAK-041 20 mg | TAK-041 40 mg
Started | 6 | 6
Completed | 5 | 5
Not Completed | 1 | 1
Not completed — PET tracer synthesis failure | 1 | 0
Not completed — Study termination | 0 | 1

BASELINE CHARACTERISTICS:
Population: The safety analysis set consisted of all participants who were enrolled and received a dose of study drug ([11C]PHNO, AMPH, or TAK-041) as part of this study.
Groups:
- TAK-041 20 mg: [11C] PHNO 180 MBq, injection, intravenously, prior to PET scan on Day 1, followed by AMPH 0.5 mg/kg, tablet, orally, once and [11C] PHNO 180 MBq, injection, intravenously, prior to PET scan post-AMPH dose on Day 2 of Confinement Period 1, followed by a 5 to 45 days of interval period, further followed by TAK-041 20 mg, suspension, orally, once, followed by AMPH 0.5 mg, tablet, orally, once and [11C] PHNO 180 MBq, injection, intravenously, prior to PET scan post-AMPH dose on Day 1 of Confinement Period 2.
- Total: Total of all reporting groups
Arm/Group | TAK-041 20 mg | TAK-041 40 mg | Total
Number analyzed (Participants) | 6 | 6 | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.2 (10.98) | 46.2 (8.16) | 39.7 (11.45)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 6 | 6 | 12
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 1 | 3
  White | 4 | 5 | 9
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Height [Mean (Standard Deviation); unit: centimeter (cm)] | 179.0 (7.46) | 177.5 (7.12) | 178.3 (7.00)
Weight [Mean (Standard Deviation); unit: kilogram (kg)] | 85.22 (4.585) | 87.90 (7.714) | 86.56 (6.210)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kilogram per square meter (kg/m^2)] | 26.65 (1.814) | 27.88 (1.375) | 27.26 (1.662)
Smoking History [Count of Participants; unit: Participants]
  Never smoked | 4 | 4 | 8
  Current smoker | 0 | 0 | 0
  Ex-smoker | 2 | 2 | 4
Alcohol History [Count of Participants; unit: Participants]
  Never drunk | 1 | 1 | 2
  Current drinker | 5 | 5 | 10
Alcohol Consumption of Less Than or Equal to (<=) 21 Units per Week [Count of Participants; unit: Participants] — Population: Alcohol consumption was assessed in the participants who were current alcohol drinker.
  Participants
    number analyzed (Participants) | 5 | 5 | 10
    (all) | 5 | 5 | 10
Caffeine History [Count of Participants; unit: Participants]
  Had caffeine consumption | 4 | 6 | 10
  Had no caffeine consumption | 2 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Change in Non-displaceable Binding Potential (BP-ND) in the TAK-041+AMPH Condition Compared to AMPH Alone
Description: The AMPH-induced change in binding potential relative to the non-displaceable component in the basal ganglia (putamen [Pu], ventral striatum [VSt]) which was the region of interest (ROI) was calculated as the percentage of reduction in specific binding from Baseline to postdose following AMPH.
Time Frame: Baseline (Day 1 of Confinement Period 1) and Day 2 post-AMPH dose in Confinement Period 1
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: percentage of reduction
Arm/Group | TAK-041 20 mg | TAK-041 40 mg
Number analyzed (Participants) | 6 | 6
percentage of reduction
  Pu | 17 (11) | 36 (8)
  VSt | 14 (14) | 23 (20)

2. Secondary Outcome: Change in BP-ND in the TAK-041+AMPH Condition Compared to AMPH Alone as a Function of the Dose of TAK-041 Administered
Description: The effect of predosing with TAK-041 on the AMPH challenge was calculated as the relative change in the percentage reduction in specific binding in ROI in the AMPH+TAK-041 condition compared to AMPH alone.
Time Frame: Baseline (Day 1 of Confinement Period 1), and Day 1 post-TAK-041 and AMPH dose in Confinement Period 2
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: percentage of reduction
Arm/Group | TAK-041 20 mg | TAK-041 40 mg
Number analyzed (Participants) | 6 | 6
percentage of reduction
  Pu | 17 (11) | 36 (8)
  Vst | 14 (14) | 23 (20)

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events are adverse events that started after the first dose of study drug and no more than 92 days after the last dose of study drug
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | TAK-041 20 mg | TAK-041 40 mg
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 0/6 | 1/6
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TAK-041 20 mg (N=6) | TAK-041 40 mg (N=6)
Pharyngitis (Infections and infestations) | 0 (0) | 1 (1)
Herpes Zoster (Infections and infestations) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Research Organization shall not publish any articles or papers nor make any presentations, nor assist any other person in publishing any articles or papers or in making any presentations relating or referring to the Study or any results, data or insights from or any data, information or materials obtained or generated in the performance of its obligations without the prior written consent of Takeda, which consent may be granted or withheld in Takeda's sole discretion.

DOCUMENTS (2):
  • Statistical Analysis Plan (2019-05-27): https://cdn.clinicaltrials.gov/large-docs/92/NCT02959892/SAP_000.pdf
  • Study Protocol (2017-02-21): https://cdn.clinicaltrials.gov/large-docs/92/NCT02959892/Prot_001.pdf